CLINICAL TRIAL: NCT01517178
Title: An Open-labelled, Randomised, Controlled, Comparative, Multi-national, Cross-over Study Investigating the Safety and Performance of a New 2-piece Ostomy Product Compared to 2-piece Standard Care Ostomy Products
Brief Title: Multi-national, Safety and Performance Study of New Ostomy Product Compared to Standard Care
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP215OC
Record Dates: First submitted 2011-06-24; First posted 2012-01-25 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Leakage; Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care base plate (Active Comparator): Standard care are the participants own product and can have several manufacture and brand names
  Interventions: Device: Standard Care base plate
- New ostomy base plate (SS) (Experimental): SS = New ostomy base plate. Due to company confidentiality the product is called SS and this is not short for any name
  Interventions: Device: New ostomy base plate (SS)

INTERVENTIONS:
Device: New ostomy base plate (SS) — The base plate is applied to the skin around the stoma and an ostomy bag is clicked onto the base plate.
  Arms: New ostomy base plate (SS)
Device: Standard Care base plate — The base plate is applied to the skin around the stoma and an ostomy bag is clicked onto the base plate.
  Arms: Standard Care base plate

SUMMARY:
The primary object of this study is to provide clinical documentation for the New base plate significantly 'reduces the degree of Leakage' under the base plate compared to Standard Care base plates.

The secondary objectives are to provide clinical documentation on several performance and safety parameters on the New base plate compared to Standard Care base plates.

The primary hypothesis is that the New base plate significantly reduces degree of leakage under the base plate compared to Standard Care base plates.

Each test period will last for two weeks. In addition to this there will be one week run-in period on New base plate. The data will be collected by investigator in the Case Report Form at the inclusion visit, cross-over visit and termination visit. Data will also be collected by the subject in a questionnaire during the two test periods.

The subjects will change their base plates on per need basis and continue with their normal changing pattern in the entire study period.

100 subjects with ileostomy will be included in the study. The subjects will be recruited from Europe including Denmark, Norway, Sweden, Iceland, Germany and France.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written Informed Consent
2. Is at least 18 years old
3. Has the mental capacity to understand the study guidelines and questionnaires
4. Has had their ileostomy for at least 3 months
5. Has an ileostomy with a diameter between 19-40 mm
6. Is currently using a flat 2-piece product with with mechanical coupling
7. Is able to change the base plate by themselves or with help from a caregiver (e.g. spouse)
8. Has experienced leakage under the base plate at least once a week over the last 2 weeks

Exclusion Criteria:

1. Is pregnant or breast-feeding
2. Currently receiving or has within the past 2 months received radio- and/or chemotherapy
3. Currently using topical steroid product on peristomal skin (injections and oral treatment are accepted)
4. Is currently using a convex base plate
5. Participating in other clinical studies or has previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Denmark (4):
  - Sygehus Sønderjylland i Aabenraa, Aabenraa
  - Bispebjerg Hospital, Copenhagen
  - Hvidovre Hospital, Hvidovre
  - Odense Universitetshospital, Odense
- France (5):
  - Hôpital Nord, Marseille
  - Hôpital Hôtel Dieu de Nantes, Nantes
  - Hôpital Lariboisière, Paris
  - CHRU La Milétrie, Poitiers
  - Hôpital de Pontchaillou, CHRU de Rennes, Rennes
- Sanitätshaus Fürst GmbH, Passau, Germany
- Landspitali University Hospital, Reykjavik, Iceland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 33 subjects were enrolled in the trial. Of these, 6 discontinued during the New ostomy base plate run-in period prior to period 1 and were excluded from the Intention-To-Treat analysis set (no performance data obtained). 27 subjects comprised the intention-to-treat population.
Groups:
- Standard Care - New Ostomy Base Plate: Subjects first test Standard Care then New ostomy base plate.
- New Ostomy Base Plate - Standard Care: Subjects first test New ostomy base plate then Standard Care.
Period: Period 1
Arm/Group | Standard Care - New Ostomy Base Plate | New Ostomy Base Plate - Standard Care
Started | 16 (One subject (who discontinued due to an adverse event) actually used New ostomy base plate.) | 11
Completed | 12 | 6
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — E.g. study termination | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Standard Care - New Ostomy Base Plate | New Ostomy Base Plate - Standard Care
Started | 11 (One subject discontinued during run-in and did not start period 2.) | 6
Completed | 5 | 4
Not Completed | 6 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — E.g. study termination | 2 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intention-to-treat Analysis Set
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Region of Enrollment [Number; unit: participants]
  France | 6
  Denmark | 19
  Iceland | 1
  Germany | 1

OUTCOME MEASURES:

1. Primary Outcome: Degree of Output Under the Base Plate (Leakage).
Description: Degree of output is measured by a 24-point leakage assessment scale (0 indicating no leakage and 24 indicating maximum leakage).
Time Frame: Each test product was assessed for 2 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Baseplates
Arm/Group | Standard Care Base Plate | New Ostomy Base Plate
Number analyzed (Participants) | 22 | 22
Number analyzed (Baseplates) | 122 | 104
units on a scale | 4.6 (3.5) | 6.5 (5.0)

ADVERSE EVENTS:
Groups:
- Standard Care Base Plate: Safety population includes subjects allocated to test period (no run-in period)
- New Ostomy Base Plate: Safety population includes subjects allocated to run-in period and test period.
Arm/Group | Standard Care Base Plate | New Ostomy Base Plate
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/30
Other Adverse Events (participants affected / at risk) | 0/21 | 13/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care Base Plate (N=21) | New Ostomy Base Plate (N=30)
Infection in parastomal prosthetic mesh (Infections and infestations) | 0 (0) | 1 (1) — Not related to the product
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care Base Plate (N=21) | New Ostomy Base Plate (N=30)
Peristomal skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) — Adverse event related or possibly related to the product
Adhesive issue (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (9) — Adverse event related to the product
Lack of effectiveness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Adverse event related to the product

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less